CLINICAL TRIAL: NCT02342639
Title: Impact of Rifaximin Therapy on Intestinal Byproducts in Chronic Kidney Disease
Brief Title: Rifaximin Therapy in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jason Stubbs, MD (Other)
Responsible Party: Sponsor-Investigator, Jason Stubbs, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00001638
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental): Participants will receive a 10-day course of Rifaximin.
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Participants will receive a 10-day course of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — 550mg pills
  Other Names: XIFAXAN®
  Arms: Rifaximin
Drug: Placebo — Placebo pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Rifaximin decreases serum and urine levels of bacterial byproducts and inflammatory markers in patients with chronic kidney disease and to evaluate changes in the bacterial content of the stool from these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease with eGFR ≤ 39 ml/min/1.73m2

Exclusion Criteria:

* Patients with normal renal function or those with less advanced kidney disease
* Inability or unwillingness to provide consent
* Patients undergoing hemodialysis or peritoneal dialysis therapy or those who have undergone organ transplant
* Patients who may be pregnant
* Hemodynamically unstable patients
* Patients with liver failure, pancreatic insufficiency, or inflammatory bowel disease
* Patients with ongoing or recent infection and those with history of C-diff infection
* Patients with abnormal bowel structure secondary to surgical or anatomic variations
* Patients on certain medications including immunosuppressants, antidiarrheal agents, bile acid sequestrants and current or recent (within the last 3 months) use of antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-06; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stubbs, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Kimber C, Zhang S, Johnson C, West RE 3rd, Prokopienko AJ, Mahnken JD, Yu AS, Hoofnagle AN, Ir D, Robertson CE, Miyazaki M, Chonchol M, Jovanovich A, Kestenbaum B, Frank DN, Nolin TD, Stubbs JR. Randomized, Placebo-Controlled Trial of Rifaximin Therapy for Lowering Gut-Derived Cardiovascular Toxins and Inflammation in CKD. Kidney360. 2020 Nov;1(11):1206-1216. doi: 10.34067/kid.0003942020. Epub 2020 Nov 25. PMID 34322673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 2015 - January 2017
Groups:
- Rifaximin: Participants will receive a 10-day course of Rifaximin 550mg PO BID.
  Rifaximin: 550mg pills
- Placebo: Participants will receive a 10-day course of placebo PO BID.
  Placebo: Placebo pill
Period: Overall Study
Arm/Group | Rifaximin | Placebo
Started | 19 | 19
Completed | 17 | 14
Not Completed | 2 | 5
Not completed — Acute illness, unrelated to study drug | 2 | 3
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rifaximin: Participants will receive a 10-day course of Rifaximin.
  Rifaximin: 550mg PO BID
- Placebo: Participants will receive a 10-day course of placebo.
  Placebo: Placebo PO BID
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Placebo | Total
Number analyzed (Participants) | 17 | 14 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13) | 65 (9) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 14 | 9 | 23
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31 (8) | 35 (9) | 33 (8)
Diagnosis of diabetes [Count of Participants; unit: Participants] — Patients with a known diagnosis of diabetes mellitus
  Participants | 7 | 11 | 18
Chronic kidney disease etiology [Count of Participants; unit: Participants]
  Diabetes | 4 | 10 | 14
  Glomerulonephritis | 1 | 0 | 1
  Hypertension | 4 | 1 | 5
  Polycystic kidney disease | 0 | 1 | 1
  Other/unknown | 8 | 2 | 10
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 27.9 (10.6) | 34.4 (14.2) | 30.8 (12.6)
Serum Trimethylamine N-oxide [Mean (Standard Deviation); unit: uM] | 18.8 (18.7) | 15.6 (11.6) | 17.3 (15.7)
Serum P-cresol sulfate [Mean (Standard Deviation); unit: ug/ml] | 18.5 (10.0) | 14.4 (4.7) | 16.7 (8.2)
Serum indoxyl sulfate [Mean (Standard Deviation); unit: ug/ml] | 3.7 (2.0) | 2.3 (0.8) | 3.1 (1.8)
Serum kynurenic acid [Mean (Standard Deviation); unit: ng/ml] | 28.1 (21.3) | 19.6 (19.0) | 24.3 (16.8)
Serum deoxycholic acid [Mean (Standard Deviation); unit: ng/ml] | 372.2 (268.3) | 609.8 (384.7) | 479.5 (342.0)
Serum C-reactive protein [Mean (Standard Deviation); unit: ug/ml] | 8.5 (22.1) | 8.2 (11.6) | 8.4 (17.9)
Serum Interleukin-6 [Mean (Standard Deviation); unit: pg/ml] | 2.1 (1.6) | 3.3 (2.6) | 2.7 (2.2)
Severity of Proteinuria [Count of Participants; unit: Participants]
  None | 6 | 6 | 12
  Mild | 4 | 4 | 8
  Moderate | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Trimethylamine N-oxide (TMAO)
Time Frame: Change from baseline to Day 11
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 17 | 14
uM | -3.9 (15.4) | 0.5 (9.5)

2. Secondary Outcome: C-reactive Protein
Time Frame: Change from baseline to Day 11
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 17 | 14
ug/ml | 6.0 (19.7) | -2.6 (5.8)

3. Secondary Outcome: Change in Serum Interleukin-6 (IL-6)
Description: post- minus pre-treatment values
Time Frame: Change from baseline to day 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 17 | 14
pg/ml | 0.3 (1.1) | 0.8 (2.1)

ADVERSE EVENTS:
Time Frame: 11 days
Arm/Group | Rifaximin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 1/17 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin (N=17) | Placebo (N=14)
Cramping/diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — GI bleeding - supra-therapeutic INR

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-08-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT02342639/Prot_SAP_ICF_000.pdf